CLINICAL TRIAL: NCT04556734
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 24-Week Study, With a 28-Week Open-Label Extension, to Assess the Safety and Efficacy of Etrasimod in Subjects With Moderate-to-Severe Alopecia Areata
Brief Title: Safety and Efficacy of Oral Etrasimod in Adult Participants With Moderate-to-Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APD334-205; C5041008 (Other: Alias Study Number)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Alopecia Areata
Keywords: T-cell-mediated autoimmune skin disorder; Alopecia areata; Alopecia; APD334; Etrasimod; Hair loss
MeSH Terms: conditions — Alopecia Areata; Alopecia | interventions — etrasimod

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Etrasimod 3 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Etrasimod — Etrasimod 3 mg (1 mg and 2 mg tablets) by mouth, once daily
  Other Names: APD334
  Arms: Etrasimod 3 mg
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of etrasimod monotherapy (2 milligrams [mg] and 3 mg) in participants with moderate-to-severe alopecia areata (AA).

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women between ≥18 and ≤70 years of age at the time of informed consent
* Moderate-to-severe alopecia areata as assessed by a SALT score of ≥25 and <95 at Screening and Day 1/Baseline.
* Current episode of hair loss for ≥6 months but <5 years
* Stable disease condition (no significant growth of hair) in the last 6 months as assessed by the Investigator
* Willing to keep the same hair style and color (eg, hair products, process, and timing for hair appointments) for the duration of the study

Key Exclusion Criteria:

* History of male or female pattern hair loss >Hamilton stage III or >Ludwig stage II
* Other types of alopecia (eg, cicatricial/scarring alopecia [including central centrifugal cicatricial alopecia], traction alopecia, or telogen effluvium) or other diseases that could cause hair loss
* Active scalp inflammation, scalp infection, scalp psoriasis, or any other scalp condition that may interfere with the SALT assessment
* Previous use of Janus kinase (JAK) inhibitor (oral or topical), including participation in clinical studies of JAK inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (39):
  - Investigate MD, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - University of California,Irvine, Irvine, California
  - Prospect Optometry, Lomita, California
  - Torrance Clinical Research Institute,Inc., Lomita, California
  - Yale Eye Center, New Haven, Connecticut
  - Yale Investigational Drug Services, New Haven, Connecticut
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Yale New Haven Hospital Department of Respiratory Care, New Haven, Connecticut
  - Advanced Sleep & Respiratory Institute, PA, Daytona Beach, Florida
  - International Eye Associates, Ormond Beach, Florida
  - Leavitt Medical Associates of Florida d/ba Ameriderm Research, Ormond Beach, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Magnante Eye Care (Ophthalmological Assessments), Lafayette, Indiana
  - Physicians Research Group (Administrative Office Location), Noblesville, Indiana
  - Physicians Research Group, West Lafayette, Indiana
  - Randall Dermatology, PC, West Lafayette, Indiana
  - Lawrence J. Green, MD LLC, Rockville, Maryland
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - NYC Retina- Manhattan, New York, New York
  - Bobby Buka MD, PC, New York, New York
  - Rochester Ophthalmological Group, Rochester, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - WDC Cosmetic and Research, PLLC, Wilmington, North Carolina
  - NW Dermatology Institute, Portland, Oregon
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Progressive Clinical Research, PA, San Antonio, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
  - PRINCIPLE RESEARCH SOLUTIONS (pulmonary function testing), Spokane, Washington
  - SPOKANE EYE CLINIC (OCT and optical exam, Spokane, Washington
- Canada (3):
  - Dermatology Research Institute, Calgary, Alberta
  - Laser Rejuvenation Clinics Edmonton D.T. Inc., Edmonton, Alberta
  - Innovaderm Research, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] King B, Mesinkovska N, Senna M, Luo X, Minkiewicz J, Selfridge A. Efficacy and safety of etrasimod in alopecia areata: A multicentre, randomized, double-blind, placebo-controlled, Phase 2 study. J Eur Acad Dermatol Venereol. 2025 Jun;39(6):1174-1184. doi: 10.1111/jdv.20605. Epub 2025 Mar 27. PMID 40145547
- [Derived] Dubinsky MC, Wu J, McDonnell A, Lazin K, Goetsch M, Branquinho D, Modesto I, Armuzzi A. Low Incidence of Macular Edema and Other Ocular Events in the Etrasimod Development Program. J Crohns Colitis. 2025 May 8;19(5):jjae173. doi: 10.1093/ecco-jcc/jjae173. PMID 39575597
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a double-blind (DB) treatment period (24 weeks) followed by an open label extension (OLE) period (28 weeks). A total of 80 participants with moderate-to-severe alopecia areata (AA) were enrolled in the DB treatment period of the study. Out of 80 participants, 65 participants entered in the subsequent OLE period.
Groups:
- DB Treatment Period: Etrasimod 2 mg: Participants who were randomized to receive etrasimod 2 milligram (mg) orally once daily for 24 weeks in DB treatment period. Participants were followed up for up to 4 weeks after last dose of study drug.
- DB Treatment Period: Etrasimod 3 mg: Participants who were randomized to receive etrasimod 2 mg orally once daily initially for Week 1 and then etrasimod 3 mg orally once daily for rest of the 23 weeks in DB treatment period. Participants were followed up for up to 4 weeks after last dose of study drug.
- DB Treatment Period: Placebo: Participants who were randomized to receive placebo matched to etrasimod orally once daily for 24 weeks in DB treatment period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period]: Participants who received etrasimod 2 mg in DB treatment period, received etrasimod 2 mg orally once daily in OLE period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period]: Participants who received placebo matched to etrasimod in DB treatment period, received etrasimod 2 mg orally once daily in OLE period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period]: Participants who received etrasimod 3 mg (also included participants whose dose was reduced from 3 mg to 2 mg due to safety issue) in DB treatment period, received etrasimod 3 mg orally once daily in OLE period either from Week 25 to Week 52 (participants who entered OLE phase on or after protocol amendment 2.0 and 2.1) or beginning after Week 25 to Week 52 in OLE period (participants who entered OLE before protocol amendment 2.0 and 2.1). Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period]: Participants who received etrasimod 2 mg in DB treatment period, received etrasimod 3 mg orally once daily in OLE period either from Week 25 to Week 52 (participants who entered OLE phase on or after protocol amendment 2.0 and 2.1) or beginning after Week 25 to Week 52 in OLE period (participants who entered OLE before protocol amendment 2.0 and 2.1). Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]: Participants received placebo matched to etrasimod in DB treatment period, received etrasimod 3 mg orally once daily in OLE period either from Week 25 to Week 52 (participants who entered OLE phase on or after protocol amendment 2.0 and 2.1) or beginning after Week 25 to Week 52 in OLE period (participants who entered OLE before protocol amendment 2.0 and 2.1). Participants were followed up for up to 4 weeks after last dose of study drug.
Period: DB Treatment Period (24 Weeks)
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]
Started | 31 | 25 | 24 | 0 | 0 | 0 | 0 | 0
Treated | 31 | 25 | 23 | 0 | 0 | 0 | 0 | 0
Completed (Completed Treatment) | 24 | 24 | 17 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 1 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: OLE Period (28 Weeks)
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]
Started | 0 | 0 | 0 | 4 (Participants who entered OLE period.) | 4 (Participants who entered OLE period.) | 24 (Participants who entered OLE period.) | 20 (Participants who entered OLE period.) | 13 (Participants who entered OLE period.)
Treated | 0 | 0 | 0 | 4 | 4 | 24 | 20 | 13
Completed (Completed treatment) | 0 | 0 | 0 | 2 | 1 | 21 | 19 | 9
Not Completed | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 4
Not completed — Not reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: DB Treatment Period randomized set included all randomized participants, irrespective of whether they received any study drug. OLE Safety set (SAF) included all participants who received at least 1 dose of study drug. Participants in DB treatment period and OLE period are not exclusive. Eligible participants from DB treatment period entered OLE period after completing treatment in DB treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period] | Total
Number analyzed (Participants) | 31 | 25 | 24 | 4 | 4 | 24 | 20 | 13 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Number Analyzed for DB treatment period and OLE Period = number of participants analyzed for reporting arms for respective period. Participants in DB treatment period and OLE period are not exclusive.
  Years
    DB Treatment Period: number analyzed (Participants) | 31 | 25 | 24 | 0 | 0 | 0 | 0 | 0 | 80
    DB Treatment Period | 36.6 (12.60) | 41.7 (16.63) | 43.4 (13.25) |  |  |  |  |  | 40.4 (14.33)
    OLE Period: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 24 | 20 | 13 | 65
    OLE Period |  |  |  | 38.0 (14.99) | 43.5 (15.67) | 42.4 (16.65) | 35.1 (12.17) | 44.8 (11.53) | 40.4 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number Analyzed for DB treatment period and OLE Period = number of participants analyzed for reporting arms for respective period. Participants in DB treatment period and OLE period are not exclusive.
  Participants
    DB Treatment Period: number analyzed (Participants) | 31 | 25 | 24 | 0 | 0 | 0 | 0 | 0 | 80
    DB Treatment Period: Female | 16 | 21 | 22 | 0 | 0 | 0 | 0 | 0 | 59
    DB Treatment Period: Male | 15 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 21
    OLE Period: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 24 | 20 | 13 | 65
    OLE Period: Female | 0 | 0 | 0 | 1 | 3 | 20 | 9 | 13 | 46
    OLE Period: Male | 0 | 0 | 0 | 3 | 1 | 4 | 11 | 0 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed for DB treatment period and OLE Period = number of participants analyzed for reporting arms for respective period. Participants in DB treatment period and OLE period are not exclusive.
  Participants
    DB Treatment Period: number analyzed (Participants) | 31 | 25 | 24 | 0 | 0 | 0 | 0 | 0 | 80
    DB Treatment Period: Hispanic or Latino | 4 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 10
    DB Treatment Period: Not Hispanic or Latino | 25 | 21 | 20 | 0 | 0 | 0 | 0 | 0 | 66
    DB Treatment Period: Unknown or Not Reported | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4
    OLE Period: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 24 | 20 | 13 | 65
    OLE Period: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 7
    OLE Period: Not Hispanic or Latino | 0 | 0 | 0 | 4 | 4 | 21 | 14 | 12 | 55
    OLE Period: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed for DB treatment period and OLE Period = number of participants analyzed for reporting arms for respective period. Participants in DB treatment period and OLE period are not exclusive.
  Participants
    DB Treatment Period: number analyzed (Participants) | 31 | 25 | 24 | 0 | 0 | 0 | 0 | 0 | 80
    DB Treatment Period: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    DB Treatment Period: Asian | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    DB Treatment Period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    DB Treatment Period: Black or African American | 2 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 11
    DB Treatment Period: White | 25 | 16 | 17 | 0 | 0 | 0 | 0 | 0 | 58
    DB Treatment Period: More than one race | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    DB Treatment Period: Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    OLE Period: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 24 | 20 | 13 | 65
    OLE Period: American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    OLE Period: Asian | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 4
    OLE Period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    OLE Period: Black or African American | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 10
    OLE Period: White | 0 | 0 | 0 | 2 | 2 | 15 | 16 | 9 | 44
    OLE Period: More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
    OLE Period: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Severity of Alopecia Tool I (SALT I) at Week 24: DB Treatment Period
Description: SALT I is a well-validated metric used to determine the degree of hair loss based on the percentage (%) of scalp surface area involved on the top (40%), back (24%), left side (18%) and right side (18%) of the scalp for AA. Investigator determines the % scalp hair loss in a given quadrant, multiply this by the total scalp area delineated by that quadrant, and sum the resultant numbers for each quadrant to give the total % scalp hair loss with a maximum score of 100. Score range from 0% (no scalp hair loss) to 100% (complete scalp hair loss), higher scores indicated more scalp hair loss. Percent change from baseline in SALT I is reported in terms of Least square mean and standard error.
Time Frame: DB Treatment Period: Baseline (before dose on Day 1), Week 24
Population: DB treatment period's full analysis set (FAS) included all randomized participants with a SALT I less than (<) 95 at baseline who received at least one dose of study drug in DB treatment period. Participants were analyzed according to the treatment they received. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change of scalp surface area
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo
Number analyzed (Participants) | 16 | 24 | 13
Percent change of scalp surface area | -13.79 (8.557) | -21.43 (6.926) | 0.35 (8.933)
Statistical Analysis 1: Comparison: DB Treatment Period: Etrasimod 2 mg vs DB Treatment Period: Placebo; Mixed model for repeated measurements (MMRM) was used for evaluation. The model included the treatment group, visit and treatment-by-visit interaction as fixed effects, disease duration and baseline SALT I score as covariates; Test type: Other — F-test; p = 0.2579, Mixed Models Analysis; LS Mean Difference = -14.14, 95% CI 2-sided [-38.933 to 10.648]
Statistical Analysis 2: Comparison: DB Treatment Period: Etrasimod 3 mg vs DB Treatment Period: Placebo; MMRM was used for evaluation. The model included the treatment group, visit and treatment-by-visit interaction as fixed effects, disease duration and baseline SALT I score as covariates; Test type: Other — F-test; p = 0.0592, Mixed Models Analysis; LS Mean Difference = -21.79, 95% CI 2-sided [-44.446 to 0.871]

2. Secondary Outcome: Change From Baseline in SALT I at Week 24: DB Treatment Period
Description: SALT I is a well-validated metric used to determine the degree of hair loss based on the percentage (%) of scalp surface area involved on the top (40%), back (24%), left side (18%) and right side (18%) of the scalp for AA. Investigator determines the % scalp hair loss in a given quadrant, multiply this by the total scalp area delineated by that quadrant, and sum the resultant numbers for each quadrant to give the total % scalp hair loss with a maximum score of 100. Score range from 0% (no scalp hair loss) to 100% (complete scalp hair loss), higher scores indicated more scalp hair loss. Change from baseline in SALT I is reported in terms of Least square mean and standard error.
Time Frame: DBT Period: Baseline, Week 24
Population: DB treatment period's FAS included all randomized participants with a SALT I <95 at baseline who received at least one dose of study drug in DB treatment period. Participants were analyzed according to the treatment they received. Here, " Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: % of scalp surface area
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo
Number analyzed (Participants) | 16 | 24 | 13
% of scalp surface area | -8.87 (4.142) | -8.62 (3.351) | 0.36 (4.314)
Statistical Analysis 1: Comparison: DB Treatment Period: Etrasimod 2 mg vs DB Treatment Period: Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other — F-test; p = 0.1283, Mixed Models Analysis; Least square (LS) Mean Difference = -9.23, 95% CI 2-sided [-21.217 to 2.748]
Statistical Analysis 2: Comparison: DB Treatment Period: Etrasimod 3 mg vs DB Treatment Period: Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other — F-test; p = 0.1057, Mixed Models Analysis; LS Mean Difference = -8.99, 95% CI 2-sided [-19.936 to 1.962]

3. Secondary Outcome: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 30%, >= 50% and >=75% Improvement From Baseline in SALT I at Week 24: DB Treatment Period
Description: SALT I is a well-validated metric used to determine the degree of hair loss based on the percentage of scalp surface area involved on the top, back, and each side of the scalp for alopecia areata (AA). Investigator determine the percent scalp hair loss in a given quadrant, multiply this by the total scalp area delineated by that quadrant, and sum the resultant numbers for each quadrant to give the total percent scalp hair loss with a maximum score of 100. Score range from 0 to 100, where 0 =no scalp hair loss to 100 = complete scalp hair loss, higher scores indicated more scalp hair loss. Percentage of participants who achieved >=30%, >=50%, >=75% improvement from baseline in SALT I at Week 24 was reported in this outcome measure.
Time Frame: DB Treatment Period: Baseline, Week 24
Population: DB treatment period's FAS included all randomized participants with a SALT I < 95 at baseline who received at least one dose of study drug in DB treatment period. Participants were analyzed according to the treatment they received. Missing data for any reason was imputed as per the non-responder imputation (NRI) method.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- DBT Period: Placebo: Participants received placebo matching to etrasimod orally once daily for 24 weeks in DBT period.
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DBT Period: Placebo
Number analyzed (Participants) | 17 | 25 | 16
Percentage of participants
  >= 30% Improvement | 23.5 [6.81 to 49.90] | 36.0 [17.97 to 57.48] | 12.5 [1.55 to 38.35]
  >= 50% Improvement | 11.8 [1.46 to 36.44] | 28.0 [12.07 to 49.39] | 12.5 [1.55 to 38.35]
  >= 75% Improvement | 5.9 [0.15 to 28.69] | 12.0 [2.55 to 31.22] | 0.000 [0.00 to 20.59]
Statistical Analysis 1: Comparison: DB Treatment Period: Etrasimod 2 mg vs DBT Period: Placebo; >= 30% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 2 mg and DB Treatment period: Placebo; Test type: Other; p = 0.4067, Cochran-Mantel-Haenszel — P-values were based on the comparison of etrasimod versus placebo; Response rate difference = 11.5, 95% CI 2-sided [-14.22 to 37.31] — Clopper-Pearson method
Statistical Analysis 2: Comparison: DB Treatment Period: Etrasimod 3 mg vs DBT Period: Placebo; >= 30% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 3 mg and DB Treatment period: Placebo; Test type: Other; p = 0.2171, Cochran-Mantel-Haenszel — P-values were based on the comparison of etrasimod versus placebo; Response rate difference = 17.5, 95% CI 2-sided [-8.23 to 43.19] — Clopper-Pearson method
Statistical Analysis 3: Comparison: DB Treatment Period: Etrasimod 2 mg vs DBT Period: Placebo; >= 50% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 2 mg and DB Treatment period: Placebo; Test type: Other; p = 0.9425, Cochran-Mantel-Haenszel — P-values were based on the comparison of etrasimod versus placebo; Response rate difference = -0.8, 95% CI 2-sided [-23.18 to 21.48] — Clopper-Pearson method
Statistical Analysis 4: Comparison: DB Treatment Period: Etrasimod 3 mg vs DBT Period: Placebo; >= 50% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 3 mg and DB Treatment period: Placebo; Test type: Other; p = 0.4959, Cochran-Mantel-Haenszel — P-values were based on the comparison of etrasimod versus placebo; Response rate difference = 8.9, 95% CI 2-sided [-15.19 to 32.94] — Clopper-Pearson method
Statistical Analysis 5: Comparison: DB Treatment Period: Etrasimod 2 mg vs DBT Period: Placebo; >= 75% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 2 mg and DB Treatment period: Placebo; Test type: Other; p = 0.3576, Cochran-Mantel-Haenszel — P-values are based on the comparison of Etrasimod versus placebo; Response rate difference = 5.6, 95% CI 2-sided [-5.39 to 16.59] — Clopper-Pearson method
Statistical Analysis 6: Comparison: DB Treatment Period: Etrasimod 3 mg vs DBT Period: Placebo; >= 75% Improvement: Response rate difference was difference in response rates between DB Treatment period: Etrasimod 3 mg and DB Treatment period: Placebo; Test type: Other; p = 0.2904, Cochran-Mantel-Haenszel — P-values were based on the comparison of etrasimod versus placebo; Response rate difference = 8.3, 95% CI 2-sided [-3.43 to 20.12] — Clopper-Pearson method

4. Other Pre Specified Outcome: Number of Participants With Adverse Events (AE): DB Treatment Period
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations based on medical significance or any diagnosis of progressive multifocal leukoencephalopathy (PML). AEs included serious AEs and all non-SAEs.
Time Frame: DB Treatment Period: From first dosing date in DB up to (before the first dosing date in OLE) or (last dosing date + 4 weeks + 3 days), whichever is earlier (maximum up to 29 weeks)
Population: DB treatment period's SAF included of all randomized participants who received at least 1 dose of study drug in DBT period. Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo
Number analyzed (Participants) | 31 | 25 | 23
Participants | 21 | 20 | 18

5. Other Pre Specified Outcome: Number of Participants With Adverse Events: OLE Period
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations based on medical significance or any diagnosis of PML. AEs included serious AEs and all non-SAEs.
Time Frame: OLE period: From first dosing date in OLE up to last dosing date + 4 weeks + 3 days (maximum up to 33 weeks)
Population: OLE period's SAF included of all participants who received at least 1 dose of study drug in the OLE Period. Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DBT]: Participants who received etrasimod 3 mg in DB treatment period, received etrasimod 3 mg orally once daily either from Week 25 to Week 52 or beginning after Week 25 to Week 52 in OLE period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period]: Participants who received etrasimod 2 mg in DB treatment period, received etrasimod 3 mg orally once daily either from Week 25 to Week 52 or beginning after Week 25 to Week 52 in OLE period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]: Participants received placebo matched to etrasimod in DB treatment period, received etrasimod 3 mg once daily either from Week 25 to Week 52 or beginning after Week 25 to Week 52 in OLE period.Participants were followed up for up to 4 weeks after last dose of study drug.
Arm/Group | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DBT] | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]
Number analyzed (Participants) | 4 | 4 | 24 | 20 | 13
Participants | 3 | 2 | 18 | 14 | 11

ADVERSE EVENTS:
Time Frame: From first dosing date up to last dosing date + 4 weeks + 3 days (maximum up to 57 weeks)
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety analysis set was evaluated.
Groups:
- OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period]: Participants who received etrasimod 2 mg in DB treatment period, received etrasimod 2 mg orally once daily in OLE period.Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period]: Participants who received placebo matched to etrasimod in DB treatment period, received etrasimod 2 mg orally once daily in OLE period.Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period]: Participants who received etrasimod 3 mg in DB treatment period, received etrasimod 3 mg orally once daily either from Week 25 to Week 52 or beginning after Week 25 to Week 52 in OLE period. Participants were followed up for up to 4 weeks after last dose of study drug.
- OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period]: Participants who received etrasimod 2 mg in DB treatment period, received etrasimod 3 mg orally once daily either from Week 25 to Week 52 or beginning after Week 25 to Week 52 in OLE period.Participants were followed up for up to 4 weeks after last dose of study drug.
Arm/Group | DB Treatment Period: Etrasimod 2 mg | DB Treatment Period: Etrasimod 3 mg | DB Treatment Period: Placebo | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period]
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/25 | 0/23 | 0/4 | 0/4 | 0/24 | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/25 | 0/23 | 1/4 | 0/4 | 1/24 | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 11/31 | 12/25 | 11/23 | 3/4 | 2/4 | 14/24 | 11/20 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Treatment Period: Etrasimod 2 mg (N=31) | DB Treatment Period: Etrasimod 3 mg (N=25) | DB Treatment Period: Placebo (N=23) | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] (N=4) | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] (N=4) | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] (N=24) | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] (N=20) | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period] (N=13)
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Treatment Period: Etrasimod 2 mg (N=31) | DB Treatment Period: Etrasimod 3 mg (N=25) | DB Treatment Period: Placebo (N=23) | OLE Period: Etrasimod 2 mg [Etrasimod 2 mg in DB Treatment Period] (N=4) | OLE Period: Etrasimod 2 mg [Placebo in DB Treatment Period] (N=4) | OLE Period: Etrasimod 3 mg [Etrasimod 3 mg in DB Treatment Period] (N=24) | OLE Period: Etrasimod 3 mg [Etrasimod 2 mg in DB Treatment Period] (N=20) | OLE Period: Etrasimod 3 mg [Placebo in DB Treatment Period] (N=13)
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 2 | 3 | 1 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 2 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyl transferase increased (Investigations) | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 4 | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fuchs' syndrome (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Retinal migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT04556734/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04556734/SAP_001.pdf